CLINICAL TRIAL: NCT00826644
Title: A Randomized Prospective Multicenter Trial of Belotecan/Cisplatin Versus Etoposide/Cisplatin in Patients With Previously Untreated, Extensive-stage Small-cell Lung Cancer
Brief Title: Trial of Belotecan/Cisplatin in Chemotherapy Naive Small Cell Lung Cancer Patient
Acronym: COMBAT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Chonnam National University Hospital (Other)
Collaborators: Chong Kun Dang Pharmaceutical (Industry)
Responsible Party: Principal Investigator, In-Jae, Oh, MD, Assistant Professor, Chonnam National University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CSCLC-0810
Record Dates: First submitted 2009-01-21; First posted 2009-01-22 (Estimated); Last update posted 2021-08-09 (Actual); Status verified 2021-08

CONDITIONS: Carcinoma, Small Cell
Keywords: Small cell lung cancer; Camptothecin; Response rate
MeSH Terms: conditions — Carcinoma, Small Cell; Small Cell Lung Carcinoma | interventions — belotecan; Etoposide; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Belotecan plus Cisplatin (Experimental)
  Interventions: Drug: Belotecan; Drug: Cisplatin
- Etoposide plus Cisplatin (Active Comparator)
  Interventions: Drug: Etoposide; Drug: Cisplatin

INTERVENTIONS:
Drug: Belotecan — Belotecan : 0.5mg/㎡/day for Day 1 to 4, repeated every 3 weeks
  Other Names: Camtobell
  Arms: Belotecan plus Cisplatin
Drug: Etoposide — Etoposide 100mg/㎡/day for Day 1 to 3, repeated every 3 weeks
  Arms: Etoposide plus Cisplatin
Drug: Cisplatin — Cisplatin 60mg/㎡/day for Day 1, repeated every 3 weeks

SUMMARY:
Belotecan (Camtobell, CKD-602, Chong Kun Dang Pharm., Korea) is a new camptothecin derivative, that exhibits anticancer effects by inhibiting topoisomerase I. The investigators will have a randomized prospective multicenter trial of Belotecan/Cisplatin versus Etoposide/Cisplatin in patients with previously untreated, extensive-stage small cell lung cancer.

Primary endpoints

* to assess Response Rate

Secondary endpoints

* to assess Overall response duration, Time to progression, Overall survival

ELIGIBILITY:
Inclusion Criteria:

* ECOG Performance status 0~2(those with performance status 2 must have been stable with no deterioration over the previous 2 weeks)
* Histologically or cytologically confirmed small cell lung cancer Patient without chemotherapy and radiotherapy
* Measurable lesion according to RECIST with at least one measurable lesion not previously irradiated, unless disease progression has been documented at that site
* Life expectancy of at least 3 months
* Provision of written informed consent

Exclusion Criteria:

* As judged by the investigator, any evidence of severe or uncontrolled systemic disease
* Serum bilirubin greater than 3 times the upper limit of reference range(ULRR)
* Aspartate aminotransferase (AST/SGOT) or alanine aminotransferase (ALT/SGPT)greater than 2.5 times ULN if no demonstrable liver metastases (or > 5 times in presence of liver metastases)
* Evidence of any other significant clinical disorder or laboratory finding that makes it undesirable for the subject to participate in the study
* Pregnancy or breast-feeding women(women of child-bearing potential). Women of childbearing potential must practice acceptable methods of birth control to prevent pregnancy
* Evidence of brain metastasis

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 147 (Actual)
Dates: Start 2009-01 (Actual); Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
To assess the response Rate of Belotecan/Cisplatin versus Etoposide/Cisplatin in patients with previously untreated, extensive-stage small cell lung cancer | two years

SECONDARY OUTCOMES:
to assess the overall response duration | two years
To assess the time to progression | two years
to assess the overall survival | two years

CONTACTS AND LOCATIONS:
Overall Officials: In-Jae Oh, M.D.,Ph.D., Principal Investigator — Chonnam National University Hospital
Locations (1):
- Chonnam National University Hwasun Hospital, Hwasun, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Oh IJ, Kim KS, Park CK, Kim YC, Lee KH, Jeong JH, Kim SY, Lee JE, Shin KC, Jang TW, Lee HK, Lee KY, Lee SY. Belotecan/cisplatin versus etoposide/cisplatin in previously untreated patients with extensive-stage small cell lung carcinoma: a multi-center randomized phase III trial. BMC Cancer. 2016 Aug 26;16(1):690. doi: 10.1186/s12885-016-2741-z. PMID 27566413